CLINICAL TRIAL: NCT04191902
Title: Educational Intervention Using SMS to Evaluate Clinical Effects and Satisfaction in Patients With Diabetes Mellitus: A Brazilian Case Study
Brief Title: Educational Intervention Using SMS to Evaluate Clinical Effects and Satisfaction in Patients With Diabetes Mellitus
Acronym: SMS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Giselle Taboada, Professor, Universidade Federal Fluminense
Other Study IDs: Diabetes Mellitus
Record Dates: First submitted 2019-11-28; First posted 2019-12-10 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Educational Problems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: control
- 2: treated
  Interventions: Behavioral: orientation

INTERVENTIONS:
Behavioral: orientation — patients will be oriented
  Groups: 2

SUMMARY:
The investigators evaluated the satisfaction of these patients with the health service and their self-care. The study included patients diagnosed with DM, respecting the established inclusion and exclusion criteria. Participants were randomized into the control group and the intervention group.

DETAILED DESCRIPTION:
Patients with diabetes mellitus (DM) have greater control over the disease when they acquire some knowledge about it. In this context, the use of technology by health professionals for nutritional guidance and self-care has shown promising results. This study aims to evaluate the impact of these educational approaches via SMS on glycemic control of patients with DM, followed at the Endocrinology Outpatient Clinic of the Antonio Pedro University Hospital (HUAP). Also, the investigators evaluated the satisfaction of these patients with the health service and their self-care. The study included patients diagnosed with DM, respecting the established inclusion and exclusion criteria. Participants were randomized into the control group and the intervention group. The patients in the intervention group received weekly SMS for six months, with dietary guidelines and DM care. Both groups answered a questionnaire at the beginning and end of the intervention, which consisted of assessing satisfaction with the health service received and their care for DM. Similarly, the investigators collected their clinical and laboratory data from medical records at the beginning and end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* diabetes

Exclusion Criteria:

* non diabetes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all patients from the ward
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-05 (Estimated); Primary Completion 2022-01-05 (Estimated); Study Completion 2022-02-15 (Estimated)

PRIMARY OUTCOMES:
differences in glycemic control | 1 year
  Evaluation of the glycemic indices

IPD SHARING:
Plan to Share IPD: No
none information will be shared